CLINICAL TRIAL: NCT05480241
Title: Impact of Exocrine Pancreatic Insufficiency Associated With Acute Pancreatitis and Pancreatic Enzyme Replacement Therapy on Gut Microbiota, Immunological Changes and Quality of Life
Brief Title: Exocrine Pancreatic Insufficiency After Acute Pancreatitis and Pancreatic Enzyme Replacement Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Unidade Local de Saúde de Coimbra, EPE (Other)
Collaborators: University of Coimbra (Other)
Responsible Party: Principal Investigator, Marta Isabel da Fonseca Gravito Soares, Principal Investigator, Unidade Local de Saúde de Coimbra, EPE
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EPInAP
Record Dates: First submitted 2022-05-22; First posted 2022-07-29 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Acute Pancreatitis; Exocrine Pancreatic Insufficiency; Gut Microbiota; Immunology
MeSH Terms: conditions — Pancreatitis; Exocrine Pancreatic Insufficiency

STUDY DESIGN:
Intervention Model Description: Double-blind randomized placebo-controlled trial for patients with EPI after acute pancreatitis for PERT and collection of stool and blood samples before and after PERT/placebo
Who Masked: Participant, Investigator
Masking Description: For evaluation the response to PERT in patients with acute pancreatitis and EPI, the study will be doubleblind (for the patient who will not know which therapy he will be taking (PERT/placebo) and for the researchers responsible for sequencing and immunological analyses) randomized placebo-controlled clinical trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pancreatic Enzyme Replacement Therapy (Experimental): Pancreatic Enzyme Replacement Therapy (PERT) 50000 Ph.U./meal + 25000 Ph.U./snack + Omeprazole 20mg once daily on fasting
  Interventions: Drug: Pancreatic Enzyme Replacement Therapy
- Placebo (Placebo Comparator): Placebo + Omeprazole 20mg once daily on fasting
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pancreatic Enzyme Replacement Therapy — Pancreatic Enzyme Replacement Therapy (PERT) 50000 Ph.U./meal + 25000 Ph.U./snack + Omeprazole 20mg once daily on fasting
  Other Names: kreon
  Arms: Pancreatic Enzyme Replacement Therapy
Drug: Placebo — Placebo + Omeprazole 20mg once daily on fasting
  Arms: Placebo

SUMMARY:
Acute pancreatitis represents an acute inflammatory process of the pancreas, which undergoes local and systemic complications, associated with non-negligible morbidity and mortality, and significant economic and quality of life impact. Even after the recovery phase, the development and persistence of sequelae from the inflammatory/necrotic process, including exocrine and endocrine pancreatic insufficiencies, are frequent. Although well documented as consequence of other pancreatic conditions, exocrine pancreatic insufficiency (EPI) after acute pancreatitis is poorly studied and probably underdiagnosed. The prevalence, diagnosis, independent risk factors and therapeutic approaches for EPI after acute pancreatitis need further investigation. Recent evidence suggests the involvement of the pancreas-intestinal axis and immunological dysfunction in several pancreatic pathologies, although their role in the development of EPI after acute pancreatitis is still scarce. Pancreatic enzyme replacement therapy (PERT) is the only treatment currently available in EPI, but the timing for start and duration of this therapy in acute pancreatitis remain to be established. This study have the following objectives: to determine the prevalence, clinical, analytical and nutritional biomarkers and duration of EPI after acute pancreatitis, as well as changes in gut microbiota and immunologic response, and quality of life in EPI and response to PERT after acute pancreatitis; and to determine the prevalence and biomarkers associated with endocrine pancreatic insufficiency following acute pancreatitis and the presence of gut dysbiosis and immunologic changes in acute pancreatitis according to its severity.

DETAILED DESCRIPTION:
Introduction: Acute pancreatitis represents an acute inflammatory process of the pancreas, which undergoes local and systemic complications, associated with non-negligible morbidity and mortality, and significant economic and quality of life impact. Even after the recovery phase, the development and persistence of sequelae from the inflammatory/necrotic process, including exocrine and endocrine pancreatic insufficiencies, are frequent. Although well documented as consequence of other pancreatic conditions, exocrine pancreatic insufficiency (EPI) after acute pancreatitis is poorly studied and probably underdiagnosed. The prevalence, diagnosis, independent risk factors and therapeutic approaches for EPI after acute pancreatitis need further investigation. Recent evidence suggests the involvement of the pancreas-intestinal axis and immunological dysfunction in several pancreatic pathologies, although their role in the development of EPI after acute pancreatitis is still scarce. Pancreatic enzyme replacement therapy (PERT) is the only treatment currently available in EPI, but the timing for start and duration of this therapy in acute pancreatitis remain to be established.

Objectives: Primary objectives: To determine the prevalence, clinical, analytical and nutritional biomarkers and duration of EPI after acute pancreatitis, as well as changes in gut microbiota and immunologic response, and quality of life in EPI and response to PERT after acute pancreatitis. Secondary objectives: To determine the prevalence and biomarkers associated with endocrine pancreatic insufficiency following acute pancreatitis and the presence of gut dysbiosis and immunologic changes in acute pancreatitis according to its severity.

Methods: Prospective longitudinal study of total of patients consecutively admitted to the Gastroenterology Department of Coimbra Hospital and University Centre with acute pancreatitis diagnosis and double-blind randomized placebo-controlled clinical trial of PERT in patients developing EPI after acute pancreatitis. This study will be conducted in 4 Phases: Phase 1 - Recruitment of patients with acute pancreatitis and stratification of them according to the severity of acute pancreatitis and development of EPI (12-month followup), diagnosed by fecal elastase-1, 13C-labeled mixed triglyceride breath test assessing exocrine pancreatic function and comparison of them with 72-hour fecal fat quantification, as gold standard; Phase 2 - Double-blind randomized placebo-controlled trial in patients with EPI after acute pancreatitis for PERT with assessment of efficacy and safety of this therapy at 1 and 6 months post-randomization; Phase 3 - Evaluation of richness, diversity and uniformity of gut microbiota by DNA sequencing using the hypervariable region of the 16S ribosomal RNA gene as a taxonomic identification marker and assessment of quality of life using SF-36 and QLC-C30-V.3 scales (validated versions for the Portuguese population) in EPI patients after acute pancreatitis, and the impact of PERT on clinical course, gut dysbiosis and quality of life of patients (at the diagnosis of acute pancreatitis, EPI and after PERT); and Phase 4 - Analysis of immunological changes through the study of cell populations by flow cytometry (CD4+, CD8+, B-cell, T-cell, natural killer cells, cells ratio) and cytokines, chemokines and growth factors by xMAP/Luminex, at the diagnosis of acute pancreatitis, EPI and after PERT.

Expected results, impact and scientific outputs: Data on the prevalence of EPI after acute pancreatitis in its different forms of severity and the role of gut dysbiosis and immunologic changes remains unclear. It's expected that an adequate and timely diagnosis of this clinical condition will allow an early start of therapy with positive impact on clinical course, immunologic and gut homeostasis, survival and quality of life. With this study we expect to obtain a prevalence of EPI at admission of 25-62%, which should decrease during followup. Alcoholic etiology, severity of acute pancreatitis and the presence of pancreatic necrosis should be positively associated with the presence of EPI after acute pancreatitis. The prevalence of endocrine pancreatic insufficiency (pre-diabetes or diabetes mellitus) should be up to 40%. Nutritional deficits (single or multiple), breath test assessing exocrine pancreatic function and fecal elastase-1 are also expected to be positively associated with the development of EPI. It's expected that patients with acute pancreatitis developing EPI will have significant changes on gut microbiota and immunologic response, and PERT and/or gut microbiota modulating therapy, including prebiotics, probiotics, symbiotics and fecal microbiota transplantation, and probably targeted immunotherapies may have a beneficial impact on all patients or groups at risk, such as EPI, severe or necrotizing acute pancreatitis by reverting gut and immunologic dysbiosis, and improving quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Definitive diagnosis of acute pancreatitis, according to revised Atlanta criteria 2012.

Exclusion Criteria:

* Age <18years
* History of allergy, hypersensitivity or contraindication to use of PERT
* Prior acute pancreatitis
* Other causes that may occur with EPI, including celiac disease, diabetic gastroparesis, chronic pancreatitis, cystic fibrosis, pancreatic neoplasia, ampulloma, somatostatinoma, somatostatin analog therapy, small bowel pathology, inflammatory bowel disease, and rare diseases associated with exocrine pancreatic insufficiency (Zollinger-Ellison syndrome, Shwachman-Diamond syndrome, Johanson-Blizzard syndrome)
* Prior gastrointestinal or pancreatic surgery or endoscopic/surgical therapy for obesity
* medication with orlistat or acarbose
* Respiratory pathology (severe chronic obstructive pulmonary disease), hepatic (Child-Pugh C cirrhosis) or biliary (obstructive jaundice) severe pathology
* Non-compliance for PERT (when indicated)
* Uncontrolled thyroid pathology
* Refusal/incapacity to give informed consent
* Follow-up period <12months after acute pancreatitis diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
When to start PERT assessed by the time, in days, between acute pancreatitis diagnosis and EPI diagnosis in patients with EPI following acute pancreatitis | Up to 12 months
  A standardized protocol will be applied for both groups differing only in drug used (PERT or placebo).
  To evaluate when to start PERT we will determine the time between acute pancreatitis diagnosis and EPI diagnosis, in days. Searching for EPI will take place up to 12 months after acute pancreatitis diagnosis.
PERT efficacy assessed by % of successful treatments in patients with EPI following acute pancreatitis | At 6 months after starting PERT
  A standardized protocol will be applied for both groups differing only in drug used (PERT or placebo). The PERT dose will be the one agreed for EPI for benign pancreatic pathologies associated with proton pump inhibitor (PPI).
  PERT efficacy will be assessed by the % of successful treatments in patients with EPI diagnosis after acute pancreatitis, using the test that was positive for EPI diagnosis (fecal elastase-1, 13 C Mixed Triglyceride Breath Test or Fecal Fat Quantitative Test). Efficacy corresponds to the normalization of exocrine pancreatic function test and will be assessed by at 6 months post-randomization. The compliance of PERT will be checked in all follow-up visits.
PERT safety assessed by adverse effects according to Medical Dictionary for Regulatory Activities in patients with EPI following acute pancreatitis | At 6 months after starting PERT
  A standardized protocol will be applied for both groups differing only in drug used (PERT or placebo). The PERT dose will be the one agreed for EPI for benign pancreatic pathologies associated with proton pump inhibitor (PPI).
  PERT safety will be evaluated with the determination of adverse effects according to Medical Dictionary for Regulatory Activities (MedDRa will be evaluated in terms of visual analogic intolerance scale (0-10) for abdominal pain and other adverse events severity in relation to the influence on activities of daily life. PERT safety will be assessed at 6 months post-randomization. The compliance of PERT will be checked in all follow-up visits.
PERT duration assessed by the time of starting PERT to normalization of exocrine pancreatic function in patients with EPI following acute pancreatitis | At 6 months after starting PERT
  A standardized protocol will be applied for both groups differing only in drug used (PERT or placebo). The PERT dose will be the one agreed for EPI for benign pancreatic pathologies associated with proton pump inhibitor (PPI).
  The duration of PERT will be evaluated determining the time, in months, between EPI diagnosis after acute pancreatitis diagnosis and the normalization of exocrine pancreatic function, determined by the normalization of positive test diagnosing EPI (fecal elastase-1, 13 C Mixed Triglyceride Breath Test or Fecal Fat Quantitative Test), using the test that was positive for EPI diagnosis.

SECONDARY OUTCOMES:
Prevalence of exocrine pancreatic insufficiency (EPI) following acute pancreatitis assessed by the proportion and percentage of patients with EPI after acute pancreatitis diagnosis | Up to 12 months
  After the recruitment of eligible patients with the first episode of acute pancreatitis, they will be stratified according to acute pancreatitis severity and EPI development. Acute pancreatitis severity will be classified into mild, moderately severe and severe cases according to the revised criteria of Atlanta 2012. The EPI diagnosis will be performed by noninvasive 13C-labeled mixed triglyceride breath test and by the non-invasive fecal elastase-1 test. At diagnosis, 72-hour fecal fat quantification will also be used as a validated indirect gold standard test.
  The prevalence of EPI will be determined by the proportion and percentage of patients with each of these complications to the total of patients with acute pancreatitis during 12-month follow-up after acute pancreatitis diagnosis. Searching for EPI will take place up to 12 months after acute pancreatitis diagnosis.
Prevalence of endocrine pancreatic insufficiency (EnPI) following acute pancreatitis assessed by the proportion and % of patients with EnPI after acute pancreatitis diagnosis | Up to 12 months
  After the recruitment of eligible patients with the first episode of acute pancreatitis, they will be stratified according to acute pancreatitis severity and EPI development. Acute pancreatitis severity will be classified into mild, moderately severe and severe cases according to the revised criteria of Atlanta 2012. Assessment of EnPI (secondary endpoint) will be defined by the development of new-onset pre-diabetes and/or diabetes mellitus - type 3 diabetes mellitus according to the diagnostic criteria of the American Diabetes Association 2019.
  The prevalence of EnPI will be determined by the proportion and percentage of patients with each of these complications to the total of patients with acute pancreatitis during 12-month follow-up after acute pancreatitis diagnosis.
Changes in gut microbiota profile using DNA sequencing of ribosomal 16S bacteria gene in acute pancreatitis, EPI following acute pancreatitis and after PERT assessed by the changes in composition and diversity of gut microbiota (OTU changes) | Change from Baseline at 6 months after starting PERT
  Analysis of gut microbiota by DNA sequencing using the hypervariable region of the ribosomal 16S bacteria gene as a taxonomic identification marker and quality of life assessment: Gut microbiota will be assessed for a number of species present (richness) and qualitative composition (diversity and uniformity) using next-generation genome sequencing techniques by an independent operator who will not know the status and therapy of EPI (PERT vs placebo). After extraction of the bacterial DNA, the sequencing of the gut microbiota by bioinformatic analysis will be performed for taxonomic identification and determination of the relative abundance of each Operational Taxonomy Units (OTU). Gut microbiota will be evaluated at baseline (acute pancreatitis diagnosis), at EPI diagnosis and 6 months after starting PERT.
Changes in Immunological profile assessed by study of cell populations in acute pancreatitis, EPI following acute pancreatitis diagnosis and after PERT | Change from Baseline at 6 months after starting PERT
  To evaluate the role of immunological response in EPI post-acute pancreatitis and PERT response, fresh peripheral blood samples will be collected and processed until obtain serum by centrifugation at 4ºC and stored at -20°C and then analyzed after the diagnosis of acute pancreatitis, after diagnosis of EPI and 6months after PERT. A standard protocol with be followed. Analysis of immunological changes: Immunological profile will be analyzed through the study of cell populations (CD4+, CD8+, B-cell, T-cell, natural killer cells, cells ratio) by multiparametric flow cytometry at acute pancreatitis diagnosis, immediately after EPI diagnosis and 6 months after PERT. This analysis will be performed by an independent operator who will not know the status and therapy of EPI (PERT vs placebo).
Changes in quality of life in patients with EPI after acute pancreatitis, EPI following acute pancreatitis and after PERT assessed by quality of life scale appropriated to this condition - SF-36 | Change from Baseline at 6 months after starting PERT
  The quality of life will be measured through the scale SF-36, validated for the Portuguese population and applicable to this pathology, that will take place after the diagnosis of acute pancreatitis, after diagnosis of EPI and 6 months after PERT. It is a 36-item questionnaire. All ofthe scales and single item scales range in score from 0 to 100. A high score for global health status/QoL represents high/healthy level of functioning and QoL.
Post-PERT changes assessed by cytokines, chemokines and growth factors in immunological profile | Change from Baseline at 6 months after starting PERT
  Fresh peripheral blood samples will be collected and processed until obtain serum by centrifugation at 4ºC and stored at -20°C and then analyzed after the diagnosis of acute pancreatitis, after diagnosis of EPI and 6months after PERT. A standard protocol with the conditions of collection, storage and transport of the different collected samples will be used. Changes from Baseline in immunological profile on cytokines, chemokines and growth factors by xMAP/Luminex at 6 months post-PERT. This analysis will be performed by an independent operator who will not know the status and therapy of EPI (PERT vs placebo).
Changes in quality of life in patients with EPI after acute pancreatitis, EPI following acute pancreatitis and after PERT assessed by quality of life scale appropriated to this condition - QLC-C30-V.3.0 | Change from Baseline at 6 months after starting PERT
  The quality of life will be measured through the scale QLC-C30-V.3.0, validated for the Portuguese population and applicable to this pathology, that will take place after the diagnosis of acute pancreatitis, after diagnosis of EPI and 6 months after PERT. It is a 30-item questionnaire. All ofthe scales and single item scales range in score from 0 to 100. A high score for functional scales and global health status/QoL represents high/healthy level of functioning and QoL. A high score for a symptom scale/item represents a high level of symptomatology or problems.

CONTACTS AND LOCATIONS:
Overall Officials: Marta Gravito-Soares, MD, Principal Investigator — Unidade Local de Saúde de Coimbra, EPE
Locations (1):
- Centro Hospitalar e Universitário de Coimbra, E.P.E., Coimbra, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lee PJ, Papachristou GI. New insights into acute pancreatitis. Nat Rev Gastroenterol Hepatol. 2019 Aug;16(8):479-496. doi: 10.1038/s41575-019-0158-2. PMID 31138897
- [Result] Roberts SE, Morrison-Rees S, John A, Williams JG, Brown TH, Samuel DG. The incidence and aetiology of acute pancreatitis across Europe. Pancreatology. 2017 Mar-Apr;17(2):155-165. doi: 10.1016/j.pan.2017.01.005. Epub 2017 Jan 19. PMID 28159463
- [Result] Xiao AY, Tan ML, Wu LM, Asrani VM, Windsor JA, Yadav D, Petrov MS. Global incidence and mortality of pancreatic diseases: a systematic review, meta-analysis, and meta-regression of population-based cohort studies. Lancet Gastroenterol Hepatol. 2016 Sep;1(1):45-55. doi: 10.1016/S2468-1253(16)30004-8. Epub 2016 Jun 28. PMID 28404111
- [Result] Banks PA, Bollen TL, Dervenis C, Gooszen HG, Johnson CD, Sarr MG, Tsiotos GG, Vege SS; Acute Pancreatitis Classification Working Group. Classification of acute pancreatitis--2012: revision of the Atlanta classification and definitions by international consensus. Gut. 2013 Jan;62(1):102-11. doi: 10.1136/gutjnl-2012-302779. Epub 2012 Oct 25. PMID 23100216
- [Result] Hollemans RA, Hallensleben NDL, Mager DJ, Kelder JC, Besselink MG, Bruno MJ, Verdonk RC, van Santvoort HC; Dutch Pancreatitis Study Group. Pancreatic exocrine insufficiency following acute pancreatitis: Systematic review and study level meta-analysis. Pancreatology. 2018 Apr;18(3):253-262. doi: 10.1016/j.pan.2018.02.009. Epub 2018 Feb 20. PMID 29482892
- [Result] Huang W, de la Iglesia-Garcia D, Baston-Rey I, Calvino-Suarez C, Larino-Noia J, Iglesias-Garcia J, Shi N, Zhang X, Cai W, Deng L, Moore D, Singh VK, Xia Q, Windsor JA, Dominguez-Munoz JE, Sutton R. Exocrine Pancreatic Insufficiency Following Acute Pancreatitis: Systematic Review and Meta-Analysis. Dig Dis Sci. 2019 Jul;64(7):1985-2005. doi: 10.1007/s10620-019-05568-9. Epub 2019 Jun 4. PMID 31161524
- [Result] Gravito-Soares M, Gravito-Soares E, Gomes D, Almeida N, Tome L. Red cell distribution width and red cell distribution width to total serum calcium ratio as major predictors of severity and mortality in acute pancreatitis. BMC Gastroenterol. 2018 Jul 5;18(1):108. doi: 10.1186/s12876-018-0834-7. PMID 29976140
- [Result] Das SL, Singh PP, Phillips AR, Murphy R, Windsor JA, Petrov MS. Newly diagnosed diabetes mellitus after acute pancreatitis: a systematic review and meta-analysis. Gut. 2014 May;63(5):818-31. doi: 10.1136/gutjnl-2013-305062. Epub 2013 Aug 8. PMID 23929695
- [Result] Ahmed Ali U, Issa Y, Hagenaars JC, Bakker OJ, van Goor H, Nieuwenhuijs VB, Bollen TL, van Ramshorst B, Witteman BJ, Brink MA, Schaapherder AF, Dejong CH, Spanier BW, Heisterkamp J, van der Harst E, van Eijck CH, Besselink MG, Gooszen HG, van Santvoort HC, Boermeester MA; Dutch Pancreatitis Study Group. Risk of Recurrent Pancreatitis and Progression to Chronic Pancreatitis After a First Episode of Acute Pancreatitis. Clin Gastroenterol Hepatol. 2016 May;14(5):738-46. doi: 10.1016/j.cgh.2015.12.040. Epub 2016 Jan 6. PMID 26772149
- [Result] Pendharkar SA, Salt K, Plank LD, Windsor JA, Petrov MS. Quality of life after acute pancreatitis: a systematic review and meta-analysis. Pancreas. 2014 Nov;43(8):1194-200. doi: 10.1097/MPA.0000000000000189. PMID 25333403
- [Result] Sankaran SJ, Xiao AY, Wu LM, Windsor JA, Forsmark CE, Petrov MS. Frequency of progression from acute to chronic pancreatitis and risk factors: a meta-analysis. Gastroenterology. 2015 Nov;149(6):1490-1500.e1. doi: 10.1053/j.gastro.2015.07.066. Epub 2015 Aug 20. PMID 26299411
- [Result] Vanga RR, Tansel A, Sidiq S, El-Serag HB, Othman MO. Diagnostic Performance of Measurement of Fecal Elastase-1 in Detection of Exocrine Pancreatic Insufficiency: Systematic Review and Meta-analysis. Clin Gastroenterol Hepatol. 2018 Aug;16(8):1220-1228.e4. doi: 10.1016/j.cgh.2018.01.027. Epub 2018 Jan 31. PMID 29374614
- [Result] Loser C, Brauer C, Aygen S, Hennemann O, Folsch UR. Comparative clinical evaluation of the 13C-mixed triglyceride breath test as an indirect pancreatic function test. Scand J Gastroenterol. 1998 Mar;33(3):327-34. doi: 10.1080/00365529850170946. PMID 9548629
- [Result] Adolph TE, Mayr L, Grabherr F, Schwarzler J, Tilg H. Pancreas-Microbiota Cross Talk in Health and Disease. Annu Rev Nutr. 2019 Aug 21;39:249-266. doi: 10.1146/annurev-nutr-082018-124306. PMID 31433743
- [Result] Zhu Y, He C, Li X, Cai Y, Hu J, Liao Y, Zhao J, Xia L, He W, Liu L, Luo C, Shu X, Cai Q, Chen Y, Lu N. Gut microbiota dysbiosis worsens the severity of acute pancreatitis in patients and mice. J Gastroenterol. 2019 Apr;54(4):347-358. doi: 10.1007/s00535-018-1529-0. Epub 2018 Dec 5. PMID 30519748
- [Result] Leal C, Almeida N. Predicting Severity in Acute Pancreatitis: A Never-Ending Quest.... GE Port J Gastroenterol. 2019 Jul;26(4):232-234. doi: 10.1159/000499680. Epub 2019 Apr 16. No abstract available. PMID 31328136
- [Result] Almeida N, Fernandes A, Casela A. Predictors of Severity and In-Hospital Mortality for Acute Pancreatitis: Is There Any Role for C-Reactive Protein Determination in the First 24 Hours? GE Port J Gastroenterol. 2015 Jul 3;22(5):187-189. doi: 10.1016/j.jpge.2015.05.004. eCollection 2015 Sep-Oct. No abstract available. PMID 28868406
- [Result] Rao SA, Kunte AR. Interleukin-6: An Early Predictive Marker for Severity of Acute Pancreatitis. Indian J Crit Care Med. 2017 Jul;21(7):424-428. doi: 10.4103/ijccm.IJCCM_478_16. PMID 28808361
- [Result] Deng LH, Hu C, Cai WH, Chen WW, Zhang XX, Shi N, Huang W, Ma Y, Jin T, Lin ZQ, Jiang K, Guo J, Yang XN, Xia Q. Plasma cytokines can help to identify the development of severe acute pancreatitis on admission. Medicine (Baltimore). 2017 Jul;96(28):e7312. doi: 10.1097/MD.0000000000007312. PMID 28700471
- [Result] Nieminen A, Maksimow M, Mentula P, Kyhala L, Kylanpaa L, Puolakkainen P, Kemppainen E, Repo H, Salmi M. Circulating cytokines in predicting development of severe acute pancreatitis. Crit Care. 2014 May 21;18(3):R104. doi: 10.1186/cc13885. PMID 24886762
- [Result] de la Iglesia-Garcia D, Huang W, Szatmary P, Baston-Rey I, Gonzalez-Lopez J, Prada-Ramallal G, Mukherjee R, Nunes QM, Dominguez-Munoz JE, Sutton R; NIHR Pancreas Biomedical Research Unit Patient Advisory Group. Efficacy of pancreatic enzyme replacement therapy in chronic pancreatitis: systematic review and meta-analysis. Gut. 2017 Aug;66(8):1354-1355. doi: 10.1136/gutjnl-2016-312529. Epub 2016 Dec 9. PMID 27941156
- [Result] Dominguez-Munoz JE. Pancreatic enzyme replacement therapy: exocrine pancreatic insufficiency after gastrointestinal surgery. HPB (Oxford). 2009 Dec;11 Suppl 3(Suppl 3):3-6. doi: 10.1111/j.1477-2574.2009.00132.x. PMID 20495625
- [Result] Kahl S, Schutte K, Glasbrenner B, Mayerle J, Simon P, Henniges F, Sander-Struckmeier S, Lerch MM, Malfertheiner P. The effect of oral pancreatic enzyme supplementation on the course and outcome of acute pancreatitis: a randomized, double-blind parallel-group study. JOP. 2014 Mar 10;15(2):165-74. doi: 10.6092/1590-8577/797. PMID 24618443
- [Result] Dominguez-Munoz JE, Nieto-Garcia L, Lopez-Diaz J, Larino-Noia J, Abdulkader I, Iglesias-Garcia J. Impact of the treatment of pancreatic exocrine insufficiency on survival of patients with unresectable pancreatic cancer: a retrospective analysis. BMC Cancer. 2018 May 5;18(1):534. doi: 10.1186/s12885-018-4439-x. PMID 29728096
- [Result] Layer P, Kashirskaya N, Gubergrits N. Contribution of pancreatic enzyme replacement therapy to survival and quality of life in patients with pancreatic exocrine insufficiency. World J Gastroenterol. 2019 May 28;25(20):2430-2441. doi: 10.3748/wjg.v25.i20.2430. PMID 31171887
- [Result] American Diabetes Association. 2. Classification and Diagnosis of Diabetes: Standards of Medical Care in Diabetes-2018. Diabetes Care. 2018 Jan;41(Suppl 1):S13-S27. doi: 10.2337/dc18-S002. PMID 29222373
- [Result] Dominguez-Munoz JE. Diagnosis and treatment of pancreatic exocrine insufficiency. Curr Opin Gastroenterol. 2018 Sep;34(5):349-354. doi: 10.1097/MOG.0000000000000459. PMID 29889111
- [Result] Ferreira PL. [Development of the Portuguese version of MOS SF-36. Part I. Cultural and linguistic adaptation]. Acta Med Port. 2000 Jan-Apr;13(1-2):55-66. Portuguese. PMID 11059056
- [Result] Pais-Ribeiro J, Pinto C, Santos C. Validation study of the portuguese version of the QLC-C30-V.3. Psic, Saúde & Doenças. 2008;9(1):89-102.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-17): https://cdn.clinicaltrials.gov/large-docs/41/NCT05480241/Prot_SAP_000.pdf
  • Informed Consent Form (2021-03-17): https://cdn.clinicaltrials.gov/large-docs/41/NCT05480241/ICF_001.pdf